CLINICAL TRIAL: NCT00643955
Title: Neuromuscular Characteristics of Individuals With Down Syndrome
Brief Title: Neuromuscular Characteristics of Individuals With Down Syndrome (DS)
Status: Terminated | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 5495
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Down Syndrome
Keywords: Evaluation of muscle strength and central activation
MeSH Terms: conditions — Down Syndrome | interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DS: Individual with Down Syndrome
  Interventions: Other: muscle strength

INTERVENTIONS:
Other: muscle strength — muscle strength

SUMMARY:
Evaluation of muscle strength and central activation of muscle in individuals with Down Syndrome

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* good health with no contraindications to exercise
* documented DS (not for control subjects)

Exclusion Criteria:

* contraindications to exercise,
* severe or profound MR
* documented atherosclerotic heart disease
* documented atlantoaxial instability
* uncorrected congenital heart disease
* implanted prosthetic device
* implanted pacemaker

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with Down Snydrome and control subjects without DS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Muscle strength Central activation ratio | One time

CONTACTS AND LOCATIONS:
Locations (1):
- IHP, Syracuse, New York, United States